CLINICAL TRIAL: NCT03761823
Title: The Pathophysiology of Post-extubation Dysphagia in ICU Patients
Brief Title: Post-extubation Dysphagia
Status: Terminated | Type: Observational
Why Stopped: Organizational issues and slow inclusion rate
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: DYSPHAGIA ICU HH17
Record Dates: First submitted 2018-02-02; First posted 2018-12-03 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2022-03

CONDITIONS: Post-extubation Dysphagia
Keywords: Flexible endoscopic evaluation of swallowing; High resolution impedance manometry; Electromyography; Intensive Care Unit

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy subjects: Healthy subjects
- Patients: Patients extubated after > 5 days of mechanical ventilation.

SUMMARY:
Mechanical ventilation is a widely used treatment on the Intensive Care Unit (ICU). Swallowing dysfunction (dysphagia) after extubation may cause aspiration, and is associated with poor outcomes: pneumonia, reintubation, a prolonged length of hospital stay and increased mortality. The exact underlying pathophysiology of post-extubation dysphagia (PED) is unknown. This exploratory pilot study is the first step that aims to fill this knowledge gap to ultimately improve current treatment and prevention of post-extubation dysphagia.

Using FEES (Flexible Endoscopic Evaluation of Swallowing), HRIM (High Resolution Impedance Manometry) and EMG (electromyography) simultaneously, 5 healthy subjects and 25 patients within 24 hours after extubation will be studied.

DETAILED DESCRIPTION:
Observational study model:

The group of healthy subjects will be recruited using posters at the local university and the internet. The healthy subjects will be studied before the group of patients to assess the feasibility and possible interactions of simultaneously recording FEES, HRIM and EMG. Then, the group of patients will be studied. They will be recruited from the Intensive Care Unit. See In- and Exclusion criteria for details.

ELIGIBILITY:
Inclusion Criteria (patients):

* age > 18 years
* informed consent
* extubated after endotracheal intubation for more than 5 days
* Richmond Agitation-Sedation Scale (RASS) between -2 and 2
* able to sit right up
* no respiratory insufficiency/failure (for this study defined as oxygen saturation (SpO2) < 92% with a minimum of 3 L nasal oxygen)

Inclusion Criteria (healthy subjects):

* age > 18 years
* informed consent

Exclusion Criteria (both patients and healthy subjects):

* pre-existing dysphagia (according to medical record and screening)
* tracheostomy or previous tracheostomy
* history of prior intubation < 3 months ago
* head/neck surgery, head/neck radiation or head/neck disease
* pre-existent esophageal disorder
* coagulopathy (thrombocytes < 50*10^9 /l, or prothrombin time (PT)/activated partial thromboplastin time (APTT) > 1.5 times the reference value, or fibrinogen < 1000 mg/l, or use of therapeutic anticoagulant drugs)
* allergy for xylometazoline (only in case its use is indicated)
* known pregnancy
* known G6PD deficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy subjects will be recruited using posters at the local university and the internet.
  Intensive care patients that will be extubated shortly.
Sampling Method: Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2019-01-22 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
The number of patients with aspiration during FEES will be assessed. | At time of measurement (within 24 hours post-extubation)

SECONDARY OUTCOMES:
Pathophysiology of PED | At time of measurement (within 24 hours post-extubation)
  The pathophysiology of PED will be determined after simultaneous measurement of FEES, HRIM and EMG. The pathophysiology will be classified into several categories: reduced pharyngeal contractility / muscular weakness, reduced upper esophageal sphincter (UES) opening/relaxation, direct oropharyngeal or laryngeal trauma of the tube, reduced laryngeal sensibility, among other categories. To enable classification, parameters obtained from FEES, HRIM and EMG will be used. FEES: presence of penetration and aspiration, residue, reduced sensibility (among others); HRIM: pharyngeal peak pressure, UES maximum admittance, intrabolus pressure (among others); EMG: duration of muscle activity (among others).
The number of adverse events will be assessed. | Participants will be followed until hospital discharge, an expected average of 28 days
Interaction of FEES on HRIM recording | At time of measurement (within 24 hours post-extubation)
  HRIM outcomes during the simultaneous recording will be compared with outcomes of recording with only HRIM in situ.
Correlation of FEES with HRIM | At time of measurement (within 24 hours post-extubation)
  The correlation of FEES outcomes, e.g. PAS and residue, with HRIM outcomes, e.g. swallow risk index and post-swallow impedance ratio.

OTHER OUTCOMES:
The number of patients that develop pneumonia will be assessed. | Participants will be followed until hospital discharge, an expected average of 28 days
  Pneumonia is defined according to the Center of Disease Control criteria.
Reintubation rate (dysphagia vs. non-dysphagia) | Participants will be followed until hospital discharge, an expected average of 28 days
  The number of patients that are reintubated during their hospital stay will be assessed.
ICU readmission rate (dysphagia vs. non-dysphagia) | Participants will be followed until hospital discharge, an expected average of 28 days
  The number of patients that are readmitted to the ICU during their hospital stay will be assessed.
Length of ICU stay (dysphagia vs. non-dysphagia) | Participants will be followed until hospital discharge, an expected average of 28 days
  Length of ICU stay will be assessed (in days).
Length of hospital stay (dysphagia vs. non-dysphagia) | Participants will be followed until hospital discharge, an expected average of 28 days
  Length of hospital stay will be assessed (in days).
ICU mortality (dysphagia vs. non-dysphagia) | Participants will be followed until hospital discharge, an expected average of 28 days
  The incidence of mortality during ICU stay will be assessed.
Hospital mortality (dysphagia vs. non-dysphagia) | Participants will be followed until hospital discharge, an expected average of 28 days
  The incidence of mortality during hospital stay will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Johannes G. van der Hoeven, prof. dr., Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboudumc, Nijmegen, Netherlands